CLINICAL TRIAL: NCT05652842
Title: Assessing the Impact of Rotational and Shift Work on Sleep, Activity, Energy Balance, and Food Choice in Adults
Acronym: SWEAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Memorial University of Newfoundland (Other)
Responsible Party: Principal Investigator, Scott Harding, Assistant Professor, Memorial University of Newfoundland
Other Study IDs: 2022.134; 20230493 (Other: Memorial University)
Record Dates: First submitted 2022-11-01; First posted 2022-12-15 (Actual); Last update posted 2022-12-15 (Actual); Status verified 2022-12

CONDITIONS: Life Style; Shift-Work; Food Preferences
Keywords: Shift work; Lifestyle; Food choice; Physical activity; Sleep
MeSH Terms: conditions — Food Preferences; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Day workers: Includes people working from 9 a.m. to 5 p.m./8 a.m. to 4 p.m. We will be recruiting 15 day workers.
  Interventions: Behavioral: Work-type
- Shift workers: Includes those involved in any arrangement of daily working hours other than the standard daylight hours, 8 a.m. - 5 p.m. It also includes on-call or casual workers. We will be recruiting 15 shift workers.
  Interventions: Behavioral: Work-type
- Rotational workers: Includes those who work on a set schedule and whose working hours are rotating on a set schedule. We do not include offshore workers here. We will be recruiting 15 rotational workers.
  Interventions: Behavioral: Work-type

INTERVENTIONS:
Behavioral: Work-type — Participants are categorized by the type of work hours they must maintain. For example, regular work hours, shift work, and rotational work.

SUMMARY:
The goal of this observational study is to compare different work schedules in adults above 30 years of age. Shift and rotational work have become increasingly common owing to the demand for 24/7 availability, especially in the province of Newfoundland, where a large cohort of workers are involved in shift working hours. There is an emerging body of evidence linking shift work with adverse health outcomes, including cardiovascular diseases, type 2 diabetes, cancer, and obesity. Short and poor-quality sleep usually results from repeated exposure to shift work, leading to disturbed circadian rhythms and energy balances. The main question this study aims to answer is the effect of shift and rotational work on physical activity, sleep and food choices in adults. Participants are required to do the following:

1. Wearing an actigraphy watch, which is very similar to any other wristwatch, for seven days to objectively record their physical activity and sleep.
2. Participants will be asked to do two 24-hour food recalls using Automated Self-Administered 24-hour (ASA24), a free dietary assessment web-based tool.
3. Fill out a few questionnaires regarding demographics, chronotype (evening or morning preference), work schedule, sleep quality, stress levels, and physical activity levels.

This is a field-based observational study collecting data both objectively and subjectively. The target population comprises 15 shift workers, 15 rotational workers and 15 daytime workers. This study will involve two visits to the lab. At the baseline, after taking informed written consent, anthropometric measurements, which include height, weight, and blood pressure, will be taken. Along with that, demographic, work schedule, and chronotype questionnaires will be filled. Participants will be instructed how to use the Actigraphy watch, ASA24, and sleep diary at home. After 7 days, participants will be asked to return to the lab to return the material. Participants will be asked to complete the physical activity, sleep quality and stress questionnaires. This study aims to monitor free-living behaviours in actual shift workers while participants are engaged in real-life work shifts.

DETAILED DESCRIPTION:
Despite the rising evidence of harmful health effects from sleep disruption caused by shift employment, society relies on it. Shift work is a broad word that refers to any work schedule that is not between the hours of 8 a.m. and 4 p.m. This study considers three groups: 1) day workers - Including people working from 9 a.m. to 5 p.m./8 a.m. to 4 p.m. 2) shift workers - Including those involved in any arrangement of daily working hours other than the standard daylight hours 8 a.m. - 5 p.m 3) rotational workers - Including those who work on set schedule and working hours are rotating on a set schedule. This study will not include offshore workers. According to the International Agency for Research on Cancer (IARC), night shift work has been classified as Group 2A, probably carcinogenic to humans, based on sufficient evidence of cancer in animals and limited evidence in humans. Shift work affects humans in many ways, mainly by disturbing the body's circadian rhythm and sleep patterns. During the night, human bodies produce melatonin and maintains a constant stream of melatonin signals that leads to sound sleeping. However, working at night puts shift workers in a circadian misalignment due to melatonin suppression. With a disturbed circadian rhythm, the different systems in the body don't function optimally. A person can struggle to fall asleep, wake up during the night, or be unable to sleep as long as they want in the morning. Another significant side effect of shift work is altered meal timing and disturbed hormonal balance. The key regulators of satiety and hunger, the hormones Leptin and Ghrelin, respectively, are driven by body's biological clock. Ghrelin stimulates appetite and decreases after meals with a reverse diurnal pattern from Leptin. Usually, these hormones work in concert to regulate feeding with meal size and time. Previous laboratory studies examining the immediate effects of circadian misalignment have demonstrated decreased Leptin levels and post-meal suppression of Ghrelin. If these results are applied to general shift workers, this may promote weight gain because of an enhanced appetite for calorie-dense foods with eating at night. Therefore, night shift workers tend to have a higher body mass index (BMI) and waist-to-hip ratio than day shift workers. Multiple epidemiological studies controlling potential confounders suggest that exposure to shift work alone can contribute to increased body weight, BMI and a higher prevalence of obesity. A long-term consequence of shift work is an increased risk of type 2 diabetes. As a result of physiological maladaptation to eating at abnormal circadian times, metabolic syndrome develops over time. Both night and rotating shifts have been associated with an elevated risk of heart disease and ischemic stroke. However, shift work and circadian irregularities do not appear to be the only factors contributing to adverse heart health outcomes but also the psychological and psychosocial stress associated with shift work.

This study's primary objective is to compare the diet patterns of day workers, shift workers and rotational workers. Previous research has shown no significant differences in the daily caloric intake of shift workers against day workers. Night workers have an enhanced preference for high-fat foods. However, in most of these studies, food intake was measured subjectively using Food Frequency Questionnaires (FFQ) and self-reported food diaries. Subjective tools may lead to inaccurate conclusions. Objective measurement of food intake in shift workers in real-life situations is required instead of a laboratory-based shift work simulation study. The international recommendation for acceptable daily macronutrient distribution for carbohydrates is 45-65%; for fats and protein, figures are 20-35% and 10-35%, respectively. This study is interested in analyzing the adherence to the daily macronutrient distribution by shift, rotational and day workers and if shift workers can achieve the recommendation for a healthy diet. The hypothesis is that shift and rotational workers would have a reduced score for vegetable, fruit and fibre intake. This research aims to study the timings and duration of food intake in workers. These factors can potentially explain the high obesity rate in shift workers and the increased risk for chronic noncommunicable diseases. Another objective is to inter compare the food intake of every worker on a working day and on a non-working day. This study is interested in seeing the caloric intake difference between the rest days and work days, frequency of eating moments, energy distribution of meals, timing of eating, and fasting intervals of workers from different categories. Considering how all these factors impact metabolic parameters like glucose tolerance and energy metabolism, evaluating these specific dietary measures is crucial.

Stress is another major factor that can influence workers' eating patterns, while only a few studies have been done to assess the impact of stress on the eating habits of shift workers. A nurse's study showed that stress significantly predicts energy and saturated fat intake. Often shift workers use food as a coping strategy for dealing with negative mood states. The objective is to compare stress levels between different worker categories and relate them to eating habits respectively.

This is a feasibility study which means data collected from this study will help determine the sample size and other factors for a large-scale intervention trial in the working cohort of Newfoundland. No previous study has been done on Newfoundland workers. This study aims to inform the design and implementation of a fully-funded trial. Data collected from this study will be used for developing hypotheses and sample sizes for future studies.

Secondary objective is to compare sleep levels in different cohorts of workers. Sleep quality is very subjective, implying that it can have different meanings for different persons. To compare sleep quality in terms of sleep duration, sleep efficiency, sleep onset time, total elapsed bedtime, and total sleep time in day workers, shift workers, and rotational workers.

To measure if shift and rotational work have any impact on the physical activity of workers. To compare the physical activity levels of different workers in terms of light/sedentary, moderate and vigorous physical activity.

It also includes collecting data to know each participant's chronotype preference. To compare this with each participant's work schedule and see if chronotype-aligned work schedules are more beneficial. Measuring objectively and subjectively each participant's physical activity and sleep quality. SWEAT study is interested in comparing both parameters' similarity and variability in the subjective and objective data. Determining the relationship between shift and rotational work and the cardiometabolic disease risk factors through the parameters we are measuring.

ELIGIBILITY:
Inclusion Criteria:

1. 30 years of age or older.
2. Should be able to wear a watch for seven days.
3. Should be working.

Exclusion Criteria:

1. Shifts less than 4.5 hours or shifts longer than 14 hours will not be considered.
2. Being pregnant.
3. Currently being breastfeeding.
4. Having a child less than 1 year old at home.
5. Travelled across time zones in the last four weeks.
6. No change in medication in the last six months for any previous ongoing medical condition (by self-reported health history).

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target study population will be recruited by advertising study directly and indirectly. We will contact local employment unions in Newfoundland to advertise our study and ask for participation, making social media accounts for the SWEAT study and advertising the study on Facebook, Instagram and Twitter. Standard passive approaches will be used, including study advertisement posters on community bulletin boards; poster distribution in public places like shopping malls, hospitals, long-term care homes, worker unions, and police departments; promotion on community radio stations, and promotion via the Memorial University Newsline.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Food Intake | Two 24-hour recalls on any day of the 7-days tracking period. Participants will be asked to complete one on working day other on non-working day, but this is not mandatory.
  Two online 24-hour food recalls using Automated Self-Administered Dietary Assessment Tool(ASA24). ASA24 is a free web-based application that allows for numerous automatically coded self-administered 24-hour recalls and dietary records for epidemiologic, interventional, behavioural, or clinical research.
Stress levels | On the second visit which is after 7 days from the first visit to the lab.
  Participants will be asked to fill the Perceived Stress Scale (PSS). It is a stress assessment instrument. It gives scores between 0-40. Higher scores means high level of stress.

SECONDARY OUTCOMES:
Sleep Measurement | Participant will be given Actigraphy watch on their first visit and will be asked to wear it for the next seven days continuously without removing. During the second visit which is after seven days, the watch will be removed by study staff.
  Sleep parameters including: total sleep time, bedtime, rise-time, sleep quality and efficiency, wake after sleep onset, sleep interruptions, posture changes using GENEActiv(Actigraphy) watch. Actigraphy is method of measuring human movement, activities and behaviours. It is normally worn on the wrist and measures temperature and environmental light as well. We are using the model GENEActiv by Activinsights Ltd, Cambs, UK.
Sleep Quality | On the second visit which is after 7 days from the first visit to the lab.
  Sleep quality will be measured using Pittsburgh Sleep Quality Index (PSQI). It is self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. It gives score between 0 and 21. Any score more than 5 is associated with poor sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Harding, Principal Investigator — Memorial University of Newfoundland
Locations (1):
- Nutrition and Lifestyle Lab, Department of Earth Sciences, Memorial University of Newfoundland, 9 Arctic Ave, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lauren S, Chen Y, Friel C, Chang BP, Shechter A. Free-Living Sleep, Food Intake, and Physical Activity in Night and Morning Shift Workers. J Am Coll Nutr. 2020 Jul;39(5):450-456. doi: 10.1080/07315724.2019.1691954. Epub 2019 Nov 19. PMID 31743081
- [Background] Siqueria K, Griep R, Rotenberg L, Silva-Costa A, Mendes da Fonseca Mde J. Weight gain and body mass index following change from daytime to night shift - a panel study with nursing professionals. Chronobiol Int. 2016;33(6):776-9. doi: 10.3109/07420528.2016.1167719. Epub 2016 May 9. PMID 27159160
- [Background] Robbins R, Quan SF, Barger LK, Czeisler CA, Fray-Witzer M, Weaver MD, Zhang Y, Redline S, Klerman EB. Self-reported sleep duration and timing: A methodological review of event definitions, context, and timeframe of related questions. Sleep Epidemiol. 2021 Dec;1:100016. doi: 10.1016/j.sleepe.2021.100016. Epub 2021 Nov 25. PMID 35761957
- [Background] Park Y, Dodd KW, Kipnis V, Thompson FE, Potischman N, Schoeller DA, Baer DJ, Midthune D, Troiano RP, Bowles H, Subar AF. Comparison of self-reported dietary intakes from the Automated Self-Administered 24-h recall, 4-d food records, and food-frequency questionnaires against recovery biomarkers. Am J Clin Nutr. 2018 Jan 1;107(1):80-93. doi: 10.1093/ajcn/nqx002. PMID 29381789
- [Background] Heath G, Dorrian J, Coates A. Associations between shift type, sleep, mood, and diet in a group of shift working nurses. Scand J Work Environ Health. 2019 Jul 1;45(4):402-412. doi: 10.5271/sjweh.3803. Epub 2019 Feb 26. PMID 30806474
- [Background] Nea FM, Pourshahidi LK, Kearney JM, Livingstone MBE, Bassul C, Corish CA. A qualitative exploration of the shift work experience: the perceived effect on eating habits, lifestyle behaviours and psychosocial wellbeing. J Public Health (Oxf). 2018 Dec 1;40(4):e482-e492. doi: 10.1093/pubmed/fdy047. PMID 29546282